CLINICAL TRIAL: NCT01106664
Title: A Double-Blind, Placebo-Controlled, Multiple Dose Escalation Study and Food Effect Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONO-7746 in Healthy Adult Subjects
Brief Title: ONO-7746 Study in Healthy Adult Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-7746POU002
Record Dates: First submitted 2010-04-13; First posted 2010-04-20 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-7746; Healthy adult subjects

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- P (Placebo Comparator)
  Interventions: Drug: ONO-7746
- E (Experimental)
  Interventions: Drug: ONO-7746

INTERVENTIONS:
Drug: ONO-7746 — 1mg, 2mg, 4mg, 8mg, 16mg, once daily for multiple-dose study; 4mg at a single dose for food effect study.
  Arms: P
Drug: ONO-7746 — 1mg, 2mg, 4mg, 8mg, 16mg once daily for multiple-dose study; 4mg at a single dose for food effect study
  Arms: E

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of NON-7746 in healthy adult subjects. The secondary objectives are to characterize the pharmacokinetic and pharmacodynamic profiles of ONO-7746 and to evaluate the food effect on the PK profile of ONO-7746 when administered with or without a meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male or female subjects (18-55 inclusive)
* Body mass index (BMI) of 19-35 kg/m2 (inclusive)
* For females, postmenopausal, non-lactating, and non-pregnant

Exclusion Criteria:

* History or presence of clinically significant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | up to 42 days
  (evaluations of physical examinations, vital signs, 12-lead ECG, slit lamp examinations, safety laboratory tests, and surveillance for adverse events)

SECONDARY OUTCOMES:
Characterization of PK and PD profiles, including platelet count changes of ONO-7746 | up to 42 days
Effect of food on ONO-7746 pharmacokinetics | up to 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Austin Clinical Site, Austin, Texas, United States